CLINICAL TRIAL: NCT01782755
Title: Probiotics: Prevention of Severe Pneumonia and Endotracheal Colonization Trial (PROSPECT): A Feasibility Clinical Trial
Acronym: PROSPECT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Technology Evaluation in the Elderly Network (TVN) (Unknown); Physician's Services Incorporated (PSI) (Unknown); Hamilton Academy of Health Science Research Organization (HAHSO) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 28012013
Record Dates: First submitted 2013-01-29; First posted 2013-02-04 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2016-03

CONDITIONS: Ventilator Associated Pneumonia (VAP); Other Infections; Antibiotic-Associated Diarrhea; C-Difficile; Duration of Mechanical Ventilation; Length of ICU Stay; Length of Hospital Stay; ICU and Hospital Mortality
Keywords: Probiotics; Ventilator Associated Pneumonia (VAP); Infection; Antibiotic-Associated Diarrhea; C-Difficile
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lactobacillus rhamnosus GG (Active Comparator): Patients allocated to the intervention group will receive 1x1010 colony forming units (CFU) of Lactobacillus rhamnosus GG (Culturelle, Locin Industries Ltd) in 1 capsule suspended in sterile water, administered through a nasogastric, nasoduodenal, percutaneous gastrostomy or percutaneous jejunal tube twice daily while patients are mechanically ventilated until 24 hours of spontaneous breathing. The first dose will be within 48 hours of intubation.
  Interventions: Drug: L. rhamnosus GG - Probiotic
- Placebo (Placebo Comparator): Patients allocated to the placebo group will receive a capsule identical in appearance to the L. rhamnosus GG capsule, but containing microcrystalline cellulose. The placebo will also be suspended in sterile water and similarly administered twice a day. When suspended in water, the placebo has identical appearance and consistency as the probiotic. The placebo will be prepared by the manufacturer of L. rhamnosus GG, Culturelle, and has been used successfully in a recent RCT in the ICU population
  Interventions: Other: Placebo - Microcrystalline Cellulose

INTERVENTIONS:
Drug: L. rhamnosus GG - Probiotic — Twice daily, patients will receive either 1x1010 colony forming units (CFU) of L. rhamnosus GG (Culturelle, Locin Industries Ltd) in 1 capsule or an identical placebo capsule
  Other Names: Culturelle Probiotic
  Arms: Lactobacillus rhamnosus GG
Other: Placebo - Microcrystalline Cellulose — Placebo capsule, twice daily (containing Microcrystalline Cellulose)
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
Probiotics are commercially available live bacteria thought to have health benefits when ingested. A literature review of probiotic studies in the intensive care unit (ICU) found that in patients who receive probiotics, there is a 25% reduction in lung infection, known as ventilator-associated pneumonia (VAP). There is also an 18% reduction in the chance of developing any infection in the ICU. However, the studies reviewed were small and not well done. Therefore, whether probiotics are really helpful or not is unclear. Before a large carefully performed study is done to evaluate the effects of probiotics in critically ill patients, a pilot trial is needed. The investigators plan to study the feasibility of such a trial in mechanically ventilated ICU patients in 11 ICUs in Ontario, investigating whether orally ingested L. rhamnosus GG (a common probiotic) prevents VAP and other infections. The 4 goals of the pilot study will be to ensure that we can successfully enrol patients; follow the protocol faithfully; make sure patients don't receive additional probiotics, and estimate how much pneumonia exists in these patients. In a separate substudy, the investigators will evaluate the effects of probiotics on lower lung infiltration with potential harmful bacteria, stool bacteria, markers of immunity called cytokines, and markers of infection called endotoxin levels. The investigators plan to enroll 150 adults admitted to ICU and receiving mechanical ventilation. Following informed consent, patients will be randomized to either L. rhamnosus GG group or an identical placebo. Twice daily, patients will receive probiotics or placebo in a feeding tube. The investigators will record all infections and other important outcomes in the ICU. This study is very important in the ongoing search for more effective strategies to prevent serious infection during critical illness. Probiotics may be an easy-to-use, readily available, inexpensive approach to help future critically ill patients around the world.

DETAILED DESCRIPTION:
Background: Probiotics are defined as live microorganisms that may confer health benefits when ingested. Meta-analysis of probiotic trials suggests a 25 % lower ventilator-associated pneumonia (VAP) and 18 % lower infection rates overall when administered to patients in the intensive care unit (ICU). However, prior trials are small, largely single center, and at high risk of bias. Before a large rigorous trial is launched, testing whether probiotics confer benefit, harm, or have no impact, a pilot trial is needed. The aim of the PROSPECT Pilot Trial is to determine the feasibility of performing a larger trial in mechanically ventilated critically ill patients investigating Lactobacillus rhamnosus GG. A priori, we determined that the feasibility of the larger trial would be based on timely recruitment, high protocol adherence, minimal contamination, and an acceptable VAP rate.

Methods/design: Patients ≥18 years old in the ICU who are anticipated to receive mechanical ventilation for ≥72 hours will be included. Patients are excluded if they are at increased risk of probiotic-associated infection, have strict enteral medication contraindications, are pregnant, previously enrolled in a related trial, or are receiving palliative care. Following informed consent, patients are randomized in variable unspecified block sizes in a fixed 1:1 ratio, stratified by ICU, and medical, surgical, or trauma admitting diagnosis. Patients receive 1 × 1010 colony forming units of L. rhamnosus GG (Culturelle, Locin Industries Ltd) or an identical placebo suspended in tap water administered twice daily via nasogastric tube in the ICU. Clinical and research staff, patients, and families are blinded.

Discussion: The primary outcomes for this pilot trial are the following: (1) recruitment success, (2) ≥90 % protocol adherence, (3) ≤5 % contamination, and (4) ~10 % VAP rate. Additional clinical outcomes are VAP, other infections, diarrhea (total, antibiotic associated, and Clostridium difficile), ICU and hospital length of stay, and mortality. The morbidity, mortality, and cost of VAP underscore the need for cost-effective prophylactic interventions. The PROSPECT Pilot Trial is the initial step toward rigorously evaluating whether probiotics decrease nosocomial infections, have no effect, or actually cause infections in critically ill patients.

Trial registration: ClinicalTrials.gov. NCT01782755

Keywords: Critically ill, Intensive care, Probiotics, Infection, Pneumonia

ELIGIBILITY:
Inclusion criteria:

1. Adults ≥18 years old in the ICU;
2. Mechanically ventilated with anticipated ventilation of ≥72 hours at enrolment.

Exclusion criteria:

1. Mechanical ventilation exceeding 72 hours at time of screening.
2. Increased risk of iatrogenic probiotic infection including specific immunocompromised populations (HIV <200 CD4 cells/μL, chronic immunosuppressive medications, prior organ or hematological transplant, neutropenia (absolute neutrophil count <500).
3. Increased risk for endovascular infection (history of rheumatic heart disease, congenital heart defect, mechanical valves, endocarditis, endovascular grafts, permanent endovascular devices such as permanent (not short-term) hemodialysis catheters, pacemakers or defibrillators).
4. Mucosal gastrointestinal tract defects (gastroesophageal or intestinal injury, including active bleeding), surgery of the esophagus, stomach, small or large bowel, liver, gallbladder, hepatobiliary tree, spleen, or pancreas within 72 hours, suspected or documented ischemic gut and severe acute pancreatitis.
5. Strict contraindication or inability to receive enteral medications.
6. Pregnancy.
7. Intent to withdraw advanced life support.
8. Enrolment in this or an ongoing related trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2013-10; Primary Completion 2014-08 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Pilot Trial - Feasibility | 90 days
  Is it feasible to perform a large RCT in mechanically ventilated critically ill patients to investigate whether orally ingested L. rhamnosus GG prevents VAP, based on successful and timely pilot trial recruitment; high adherence to protocol; minimal contamination; and an acceptable VAP rate?

CONTACTS AND LOCATIONS:
Overall Officials: Deborah J Cook, MD, Principal Investigator — McMaster University
Locations (14):
- United States (2):
  - Mayo Clinic, Rochester, Minnesota
  - St. John's Mercy Medical Center, St Louis, Missouri
- Canada (12):
  - Vancouver General Hospital, Vancouver, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia
  - Vancouver Island Health Authority, Victoria, British Columbia
  - Hamilton Health Science - Hamilton General Hospital, Hamilton, Ontario
  - St Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Hamilton Health Science - Juravinski Hospital, Hamilton, Ontario
  - Ottawa Hospital Research Institute - Civic Campus, Ottawa, Ontario
  - Ottawa Research Institute - General Hospital, Ottawa, Ontario
  - St Michael's Hospital, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - University Health Network - Toronto Western Hospital, Toronto, Ontario
  - Hopital de l'Enfant Jesus, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lau VI, Xie F, Fowler RA, Rochwerg B, Johnstone J, Lauzier F, Marshall JC, Basmaji J, Henderson W, Khwaja K, Loubani O, Niven DJ, Zarychanski R, Arabi YM, Cartin-Ceba R, Thabane L, Heels-Ansdell D, Cook DJ. Health economic evaluation alongside the Probiotics to Prevent Severe Pneumonia and Endotracheal Colonization Trial (E-PROSPECT): a cost-effectiveness analysis. Can J Anaesth. 2022 Dec;69(12):1515-1526. doi: 10.1007/s12630-022-02335-9. Epub 2022 Oct 26. PMID 36289153
- [Derived] Lau VI, Cook DJ, Fowler R, Rochwerg B, Johnstone J, Lauzier F, Marshall JC, Basmaji J, Heels-Ansdell D, Thabane L, Xie F; PROSPECT Collaborators. Economic evaluation alongside the Probiotics to Prevent Severe Pneumonia and Endotracheal Colonization Trial (E-PROSPECT): study protocol. BMJ Open. 2020 Jun 28;10(6):e036047. doi: 10.1136/bmjopen-2019-036047. PMID 32595159
- [Derived] Lamarche D, Johnstone J, Zytaruk N, Clarke F, Hand L, Loukov D, Szamosi JC, Rossi L, Schenck LP, Verschoor CP, McDonald E, Meade MO, Marshall JC, Bowdish DME, Karachi T, Heels-Ansdell D, Cook DJ, Surette MG; PROSPECT Investigators; Canadian Critical Care Trials Group; Canadian Critical Care Translational Biology Group. Microbial dysbiosis and mortality during mechanical ventilation: a prospective observational study. Respir Res. 2018 Dec 7;19(1):245. doi: 10.1186/s12931-018-0950-5. PMID 30526610
- [Derived] Johnstone J, Meade M, Marshall J, Heyland DK, Surette MG, Bowdish DM, Lauzier F, Thebane L, Cook DJ; PROSPECT Investigators and the Canadian Critical Care Trials Group. Probiotics: Prevention of Severe Pneumonia and Endotracheal Colonization Trial-PROSPECT: protocol for a feasibility randomized pilot trial. Pilot Feasibility Stud. 2015 May 24;1:19. doi: 10.1186/s40814-015-0013-3. eCollection 2015. PMID 27965798
- [Derived] Cook DJ, Johnstone J, Marshall JC, Lauzier F, Thabane L, Mehta S, Dodek PM, McIntyre L, Pagliarello J, Henderson W, Taylor RW, Cartin-Ceba R, Golan E, Herridge M, Wood G, Ovakim D, Karachi T, Surette MG, Bowdish DM, Lamarche D, Verschoor CP, Duan EH, Heels-Ansdell D, Arabi Y, Meade M; PROSPECT Investigators and the Canadian Critical Care Trials Group. Probiotics: Prevention of Severe Pneumonia and Endotracheal Colonization Trial-PROSPECT: a pilot trial. Trials. 2016 Aug 2;17:377. doi: 10.1186/s13063-016-1495-x. PMID 27480757
- See also: PROSPECT Trial — http://prospecttrial.com/